CLINICAL TRIAL: NCT03370003
Title: Operational Experience With Non-routine Use of Antibiotics in the Treatment of Severe Uncomplicated Acute Malnutrition in Children
Brief Title: Non-routine Use of Antibiotics (Amoxi-light)
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Médecins Sans Frontières, France (Other)
Responsible Party: Sponsor
Other Study IDs: NE-914
Record Dates: First submitted 2017-11-21; First posted 2017-12-12 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard medical care — All children will receive nutritional treatment and standard medical care in accordance with the nutritional guidelines of the national protocol, with the exception of the routine distribution of antibiotics.

SUMMARY:
To evaluate, in routine operational settings of treatment of uncomplicated Severe Acute Malnutrition (SAM) in children aged 6-59 months, the risk of nutritional recovery and hospitalization with non-routine use of amoxicillin compared to the risk achieved with systematic use of antibiotics.

DETAILED DESCRIPTION:
Upon admission, all children will receive nutritional treatment and standard medical care in accordance with the nutritional guidelines of the national protocol, with the exception of the routine distribution of antibiotics. Antibiotics will be provided at admission and during follow-up only if clinically justified. The results of the program (ie, nutritional recovery, hospitalization, death and abandonment) will be monitored in all children aged 6 to 59 months admitted for outpatient therapy in 2 outpatient treatment sites in the Madarounfa health district in Niger.

To ensure that the children included in the study receive appropriate care, the study will ask the children's leaders to return to the clinic for medical surveillance in the event of a clinical complication. Program staff will facilitate appropriate management, including prescription of antibiotics if clinically justified, and transfer to hospital of all children in need of close supervision and / or comprehensive medical management.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months
* Direct admission for the treatment of uncomplicated SAM (MUAC <115 mm or PTZ <-3 and / or presence of Grade + or ++ nutritional edema and moderate or good appetite with absence of medical complications)
* Signed Informed Consent

Exclusion Criteria:

* No Informed Consent given
* Not directly admitted for the treatment of uncomplicated SAM at the CRENAS (Center for Outpatient Nutritional Rehabilitation for Malnutrition) of the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children from 6 to 59 months admitted directly for the treatment of uncomplicated SAM(MUAC <115 mm or PTZ <-3 and / or presence of nutritional edema grade + or + + and moderate or good appetite with no medical complications) in the 2 CRENAS chosen as study sites during the inclusion period of the study. A "direct admission" is defined as an admission without reference from CRENI (intensive nutritional recovery and education centres) to CRENAS. Readmission cases, that is, children admitted to the nutritional program in the last 3 months, and references from the Center for Ambulatory Nutritional Recovery for Moderates (CRENAM) remain eligible for inclusion of the study without prejudice and without notation at the previous admission.
Sampling Method: Non-Probability Sample
Enrollment: 2876 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of nutritional recovery | Through study participation, no more than 2 months after follow-up of the last participant
  Primary outcome will be measured in the field of nutrition, hospitalization, death and abandonment in the observation site (s) with that observed in 3 comparison groups:
  1. Children receiving amoxicillin and placebo in the randomized trial conducted by MSF (2012-2014)
  2. Children receiving amoxicillin in MSF program sites not selected for study in Madarounfa (2016)
  3. Children receiving amoxicillin at selected sites from the previous year (2015)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca GRAIS, PhD, Study Director — Epicentre

IPD SHARING:
Plan to Share IPD: No
The results of the study will be regularly communicated to all partners. A scientific article will be prepared and presented to the reading committee of a specialized journal, as well as to international symposia, in order to allow wide dissemination to the scientific community.
  MSF standard policy on data sharing will apply.